CLINICAL TRIAL: NCT06922279
Title: First Line gastroeSOphageal metastatiC canceR primAry and disTant (if Oligometastatic) lEsions-directed Radiotherapy, a Multicentric, Phase III, Randomized Controlled Trial
Acronym: SOCRATE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, CELLINI FRANCESCO, Clinical Professor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0001634/24
Record Dates: First submitted 2025-03-26; First posted 2025-04-10 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-03

CONDITIONS: Gastroesophageal Cancer (GC)
Keywords: Gastroesophageal cancer; metastatic gastroesophageal cancer
MeSH Terms: interventions — Radiotherapy; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard systemic therapy without RT/SBRT combination (Other): The patients will go to standard therapy (chemotherapy treatment with carboplatin-taxol or with drugs that the oncologist that the oncologist considers most useful.) without RT/SBRT combination
  Interventions: Drug: Standard systemic therapy (chemotherapy)
- Standard systemic therapy with RT/SBRT combination (Experimental): Standard systemic therapy (chemotherapy treatment with carboplatin-taxol or with drugs that the oncologist considers most useful) + combination of RT on the primary gastroesophageal Gross Tumor Volume (GTV) + SBRT on each of the distal lesions for oligometastatic or limited metastatic spread patients (to be delivered prior to initiation of systemic therapy).
  Interventions: Radiation: Radiation Therapy + standard sistemic therapy (chemoteraphy)

INTERVENTIONS:
Radiation: Radiation Therapy + standard sistemic therapy (chemoteraphy) — Standard systemic therapy (chemotherapy treatment with carboplatin-taxol or with drugs that the oncologist considers most useful) + combination of RT on the primary gastroesophageal Gross Tumor Volume (GTV) + SBRT on each of the distal lesions for oligometastatic or limited metastatic spread patients (to be delivered prior to initiation of systemic therapy).
  Other Names: SBRT
  Arms: Standard systemic therapy with RT/SBRT combination
Drug: Standard systemic therapy (chemotherapy) — The patients will go to standard therapy (chemotherapy treatment with carboplatin-taxol or with drugs that the oncologist that the oncologist considers most useful.) without RT/SBRT combination
  Other Names: sistemic therapy; No radiation; standard
  Arms: Standard systemic therapy without RT/SBRT combination

SUMMARY:
The aim of the study is to evaluate the efficacy of radiotherapy on the primary site of gastroesophageal cancer and extracranial stereotactic radiotherapy on metastases before the use of standard systemic therapy, in cases of limited disease burden (in the experimental group), compared to the standard group, which does not receive radiotherapy. This prospective, multicenter, randomized trial aims to evaluate the efficacy of the unconventional approach versus the conventional one in increasing the percentage of asymptomatic patients due to the direct effect of the primary tumor or metastases. "Randomized" means that the assignment to one of the treatment groups mentioned above will be random, not influenced by the physician or the patient's condition. Therefore, your participation in either of the two treatments under study will be assigned randomly and not predetermined. This randomness is crucial for a proper analysis of the results at the end of the study, which will help clarify whether there are differences between the two proposed treatments. This also means that you may not receive direct benefits from participating in this study, as it is a research study.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with gastroesophageal cancer (i.e.: esophagus, gastroesophageal junction, stomach), for both major squamous cell (SCC) and adenocarcinomatous (ADK) histologies, metastatic, candidate for first-line standard systemic treatment; either newly diagnosed in metastatic stage or first progression to metastasis.
* Obtaining informed consent.
* Patients >18 years of age
* ECOG 0-2
* Performance of imaging (CT with mdc, MRI with mdc, CT-PET with appropriate tracer) adequate for baseline local and systemic staging and likely to be similarly repeatable at 6 and 12 months after randomization
* Confirmation at the time of randomization, by the Radiation Therapy Center, that all potentially planned treatments can be performed for the patient (if enrolled in experimental arm) within a maximum of 25 days total before referral to the Medical Oncology Center for systemic therapy

Exclusion Criteria:

* Metastatic picture of line following the first
* Technical or organizational inability to the eventual deadline for radiation treatments within 25 days of randomization
* Inability to express independent consent to treatments
* Pregnancy
* Patient in hospice or with prognosis < 6 months
* Predicted unavailability for follow-up at 6 months
* Absence of adequate or likely non-repeatable pretreatment imaging study at 6 and 12 months
* Previous radiation therapy
* Previous radiometabolic therapy
* Inability to maintain treatment position for SBRT
* Symptomatic emergent or other presentation precluding study development as planned (e.g., epidural compression of the spinal cord or cauda equina)
* Previous chemotherapy, immunotherapy or target therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2024-11-30 (Actual); Primary Completion 2029-10-30 (Estimated); Study Completion 2029-11-30 (Estimated)

PRIMARY OUTCOMES:
Disappearance of symptoms | From the week after the treatment up to 12 months after
  Percentage difference in the rate of patients with symptom (from primary tumor or metastasis) developed within the first 6 months.

SECONDARY OUTCOMES:
Pain level | From the week after the treatment up to 12 months after
  Level of metastasis-associated or primary pain (presence/absence, level and response) at 6 months
Radiotherapy use | From the week after the treatment up to 12 months after
  Rate of recourse to Radiotherapy for pain, obstruction, bleeding or other symptom referable to the primary at 6 months from randomization (and not present at randomization)

CONTACTS AND LOCATIONS:
Locations (1):
- Policlinico Universitario Agostino Gemelli IRCSS, Rome, RM, Italy

IPD SHARING:
Plan to Share IPD: Undecided